CLINICAL TRIAL: NCT05777707
Title: Neoadjuvant Therapy of PD-1 Blockade Combined With Chemotherapy for Locally Advanced Esophageal Carcinoma
Brief Title: Neoadjuvant Therapy of PD-1 Blockade Combined With Chemotherapy for Esophageal Carcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BeijingHF
Record Dates: First submitted 2023-01-30; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-01

CONDITIONS: Esophageal Carcinoma; Neoadjuvant Immunotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Immune Checkpoint Inhibitors; Carboplatin; nedaplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant PD-1 Blockade Plus Chemotherapy (Experimental): PD-1 blockade, 200 mg, IV., every 3 weeks, 2-3 cycles； Albumin paclitaxel, 300 mg/m2, IV., every 3 weeks, 2-3 cycles； Carboplatin/Nedaplatin, area under the curve = 5, IV., every 3 weeks, 2-3 cycles.
  Interventions: Drug: PD-1 blockade; Drug: Albumin paclitaxel; Drug: Carboplatin/Nedaplatin

INTERVENTIONS:
Drug: PD-1 blockade — PD-1 blockade (Sintilimab/Camrelizumab/Toripalimab/Tislelizumab), 200 mg, IV., every 3 weeks, 2-3 cycles.
Drug: Albumin paclitaxel — Albumin paclitaxel, 300 mg/m2, IV., every 3 weeks, 2-3 cycles.
Drug: Carboplatin/Nedaplatin — Carboplatin/Nedaplatin, area under the curve = 5, IV., every 3 weeks, 2-3 cycles.

SUMMARY:
This prospective study aims to clarify the clinical efficacy and survival prognosis of neoadjuvant immune checkpoint inhibitor (ICI) combined with chemotherapy for esophageal cancer. It also explores predictive biomarkers and potential therapeutic targets for locally advanced esophageal cancer based on plasma metabolomics and peripheral blood immune cell clustering analysis. Each patient received 2-3 cycles of neoadjuvant immunotherapy with programmed cell death 1 (PD-1) blockade in combination with albumin paclitaxel and platinum. Exploratory analysis of plasma metabolomics combined with peripheral blood subsets of immune cells can reveal biomarkers that predict the efficacy and prognosis of patients undergoing neoadjuvant immunotherapy for locally advanced esophageal cancer, which also provide new ideas for the selection of immune adjuvants and therapeutic targets in ICIs combination therapy strategies.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years and ≤89 years;
2. pathological histological examination confirmed the diagnosis of esophageal squamous cell carcinoma and esophageal adenocarcinoma;
3. clinical stage II-IVA;
4. adequate organ function;
5. no previous chemotherapy or radiotherapy;
6. voluntarily signed informed consent.

Exclusion Criteria:

1. the presence of concurrent malignancies that interfere with the prognosis of esophageal cancer;
2. patients with immunodeficiency or autoimmune diseases that seriously affect the body's immune system, such as those who test positive for HIV;
3. patients undergoing systemic corticosteroid or other immunosuppressive treatments;
4. patients with a history of allergy to the components of this test drug.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Estimated)
Dates: Start 2020-10-29 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 24 months
  Disease-free survival was defined as the time from randomization until the first documented disease recurrence or death due to any cause.

SECONDARY OUTCOMES:
Pathologic complete remission (PCR) | 4 weeks after surgery
  Primary tumor or lymph node surgery specimen pathological examination without residual tumor cell.
Major Pathologic Response (MPR) | 4 weeks after surgery
  MPR was defined as the presence of viable tumor cells≤10% in the resected tumor specimen.
Overall survival (OS) | 24 months
  Overall survival was defined as the time from randomization grouping to the time of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Qin li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.